CLINICAL TRIAL: NCT01879410
Title: DB2114951: A Randomized, Multi-center, Double-blind, Double-dummy, Parallel Group Study to Evaluate the Efficacy Umeclidinium/Vilanterol Compared With Fluticasone Propionate/Salmeterol Over 12 Weeks in Subjects With COPD
Brief Title: A Study to Compare the Efficacy and Safety of Umeclidinium/Vilanterol With Fluticasone Propionate/Salmeterol in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114951
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK573719; lung function; salmeterol (SAL); umeclidinium bromide (UMEC); GW642444; Chronic obstructive pulmonary disease; Novel Dry Powder Inhaler (NDPI); fluticasone propionate (FP); vilanterol (VI)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- UMEC/ VI via NDPI + placebo ACCUHALER/DISKUS arm (Experimental): Subjects will receive one inhalation of UMEC/VI 62.5/25 mcg once-daily in the morning via the NDPI and one inhalation of placebo in the morning and evening via ACCUHALER/DISKUS inhaler
  Interventions: Drug: UMEC/VI Inhalation Powder 62.5/25 mcg via NDPI; Drug: Placebo DISKUS
- FSC via ACCUHALER/DISKUS + placebo NDPI arm (Active Comparator): Subjects will receive one inhalation of FSC 250/50 mcg in the morning and evening via ACCUHALER/DISKUS inhaler and one inhalation of placebo administered once-daily in the morning via NDPI
  Interventions: Drug: FSC Inhalation Powder 250/50 mcg via ACCUHALER/DISKUS; Drug: Placebo NDPI

INTERVENTIONS:
Drug: UMEC/VI Inhalation Powder 62.5/25 mcg via NDPI — The drug is administered via NDPI as one inhalation once daily in the morning. NDPI has two strips, each containing 30 blisters of medication. The first strip has UMEC blended with lactose and magnesium stearate in the form of dry white powder with a dosage of 62.5 mcg per blister and the second strip has VI blended with lactose and magnesium stearate in the form of dry white powder with a dosage of 25 mcg per blister.
  Arms: UMEC/ VI via NDPI + placebo ACCUHALER/DISKUS arm
Drug: FSC Inhalation Powder 250/50 mcg via ACCUHALER/DISKUS — The drug is administered via ACCUHALER/DISKUS inhaler as one inhalation each morning and evening. The inhaler contains a single strip with 60 blisters of medication. The strip has 250 mcg of fluticasone propionate and 50 mcg of salmeterol per blister in the form of dry white powder.
  Arms: FSC via ACCUHALER/DISKUS + placebo NDPI arm
Drug: Placebo DISKUS — Placebo is administered via ACCUHALER/DISKUS inhaler as one inhalation each morning and evening. The inhaler contains 1 strip with 60 blisters of placebo in the form of dry white powder.
  Arms: UMEC/ VI via NDPI + placebo ACCUHALER/DISKUS arm
Drug: Placebo NDPI — Placebo is administered via NDPI as one inhalation once daily in the morning. The inhaler contains 2 strips with 30 blisters of placebo per strip in the form of dry white powder.
  Arms: FSC via ACCUHALER/DISKUS + placebo NDPI arm

SUMMARY:
Umeclidinium/vilanterol (UMEC/VI) is a combination product under development that is used for the treatment of airflow obstruction in patients with COPD. Fluticasone propionate/salmeterol (FSC) is an approved drug that is already in use for the treatment of COPD. This is a multicenter, randomized, double-blind, double-dummy, parallel group study to evaluate the efficacy and safety of UMEC/VI 62.5/25 microgram [mcg] once daily administered via Novel Dry Powder Inhaler (NDPI) compared with fluticasone propionate /salmeterol (FSC) 250/50 mcg twice-daily when administered via ACCUHALER/DISKUS inhaler over a treatment period of 12 weeks in subjects with COPD. Eligible subjects will be equally randomized to UMEC/VI 62.5/25 mcg or FSC 250/50 mcg for 12 weeks. A safety follow-up assessment will be conducted approximately 7 days after the end of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: Subjects 40 years of age or older at Visit 1.
* Gender: Male or female subjects. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Or if of child bearing potential, has a negative pregnancy test at screening, and agrees to one of the acceptable contraceptive methods mentioned in the protocol used consistently and correctly:
* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society as follows: COPD is a preventable and treatable disease state characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.
* Smoking history: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years [number of pack years = (number of cigarettes per day/20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack year history.
* Severity of disease: A pre and post-salbutamol FEV1/FVC ratio of <0.70 and a post-salbutamol FEV1 of >=30% and <=70% of predicted normal values calculated using National Health and Nutrition Examination Survey (NHANES) III reference equations at Visit 1.
* Dyspnea: A score of >=2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Visit 1.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject, who, in the opinion of the investigator, has any other significant respiratory condition in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease. Inactive tuberculosis in more than one lobe is exclusionary. Allergic rhinitis is not exclusionary.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, corticosteroid, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
* Hospitalization: Hospitalization for pneumonia within 12 weeks prior to Visit 1.
* History of COPD Exacerbation: A documented history of at least one COPD exacerbation in the 12 months prior to Visit 1 that required either oral corticosteroids, antibiotics, and/or hospitalization. Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnea, sputum volume, or sputum purulence.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* 12-Lead electrocardiogram (ECG): An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility.
* Medication Prior to Spirometry: Unable to withhold salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids - 12 weeks, Systemic, oral or parenteral corticosteroids - 6 weeks, Antibiotics (for lower respiratory tract infection) - 6 weeks, Cytochrome P450 3A4 strong inhibitors - 6 weeks, Herbal medications potentially containing oral or systemic steroids - 6 weeks, Inhaled corticosteroids (ICS) - 30 days, Long-acting beta2-agonist (LABA)/ICS combination products - 30 days, Phosphodiesterase 4 (PDE4) inhibitors (e.g., roflumilast) - 14 days, Inhaled long-acting anticholinergics - 7 days, Olodaterol and Indacaterol - 10days, Theophyllines - 48 hours, Oral leukotriene inhibitors (zafirlukast, montelukast, zileuton) - 48 hours, Oral beta2-agonists Long-acting-48 hours/Short-acting - 12 hours, Inhaled long acting beta2-agonists (LABA, e.g., salmeterol, formoterol, indacaterol) - 48 hours, Inhaled sodium cromoglycate or nedocromil sodium - 24 hours, Inhaled short acting beta2-agonists - 4 hours, Inhaled short-acting anticholinergics - 4 hours, Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products - 4 hours, Any other investigational medication - 30 days or within 5 drug half-lives (whichever is longer).
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <=12 hours per day) is not ex-clusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* Inability to read: A subject will not be eligible for the study if in the opinion of the investigator the subject cannot read.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2013-06-13; Primary Completion 2014-01-01 (Actual); Study Completion 2014-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- United States (15):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Renton, Washington
- Chile (6):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Talca, Región Metro de Santiago
  - GSK Investigational Site, Talcahuano
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México DF
  - GSK Investigational Site, Oaxaca City
- Norway (6):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Bodø
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Kløfta
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Trondheim
- Romania (7):
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Comuna Alexandru Cel Bun
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Focşani
- Russia (18):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Chita
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Vladimir
  - GSK Investigational Site, Vladivostok
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- South Africa (8):
  - GSK Investigational Site, Meyerspark, Gauteng
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Die Wilgers
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Reiger Park
  - GSK Investigational Site, Somerset West

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Donohue JF, Worsley S, Zhu CQ, Hardaker L, Church A. Improvements in lung function with umeclidinium/vilanterol versus fluticasone propionate/salmeterol in patients with moderate-to-severe COPD and infrequent exacerbations. Respir Med. 2015 Jul;109(7):870-81. doi: 10.1016/j.rmed.2015.04.018. Epub 2015 May 8. PMID 26006754
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 700 participants representing the enrolled participants, were randomized to study treatment. Of these, 697 comprised the Intent-to-Treat Population (participants randomized to treatment who received >=1 dose of randomized study medication in the treatment period).
Groups:
- UMEC/VI 62.5/25 µg: Participants received umeclidinium bromide/vilanterol (UMEC/VI) 62.5/25 micrograms (µg)) once daily (QD) in the morning via a dry powder inhaler (DPI) and placebo in the morning and evening via a separate DPI for 12 weeks.
- FSC 250/50 µg: Participants received fluticasone propionate/salmeterol (FSC) 250/50 µg twice daily (BID) in the morning and evening via a DPI and placebo in the morning via a separate DPI for 12 weeks.
Period: Overall Study
Arm/Group | UMEC/VI 62.5/25 µg | FSC 250/50 µg
Started | 350 | 350
Intent-to-Treat Population | 349 | 348
Completed | 326 | 312
Not Completed | 24 | 38
Not completed — Adverse Event | 9 | 14
Not completed — Lack of Efficacy | 4 | 6
Not completed — Protocol Violation | 1 | 7
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Randomised in Error | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- UMEC/VI 62.5/25 mcg: Participants received UMEC/VI 62.5/25 µg QD in the morning via a DPI and placebo in the morning and evening via a separate DPI for 12 weeks.
- FSC 250/50 mcg: Participants received FSC 250/50 µg BID in the morning and evening via a DPI and placebo in the morning via a separate DPI for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | UMEC/VI 62.5/25 mcg | FSC 250/50 mcg | Total
Number analyzed (Participants) | 349 | 348 | 697
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (8.57) | 64.0 (8.53) | 63.6 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 84 | 169
  Male | 264 | 264 | 528
Race/Ethnicity, Customized [Number; unit: Particpants]
  African American/African Heritage | 18 | 13 | 31
  American Indian or Alaska Native | 7 | 2 | 9
  Asian | 4 | 2 | 6
  White | 317 | 326 | 643
  American Indian or Alaska Native & White | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in 0 to 24 Hour Weighted Mean Forced Expiratory Volume Over 1 Second (FEV1) at Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean was calculated from the pre-dose FEV1 and post-dose FEV1 measurements at 5 and 15 minutes and 1, 3, 6, 9, 12 hours (pre-evening dose), 13, 15, 18, 23, and 24 hours after the morning dose. Baseline is defined as the mean of the assessments made 30 and 5 minutes (min) pre-dose on treatment Day 1. Analysis was performed using an analysis of covariance model with covariates of baseline FEV1 (mean of the two assessments made 30 mins and 5 mins pre-dose on Day 1), smoking status, and treatment. Change from baseline was calculated as the value at Day 84 minus the value at Baseline.
Time Frame: Baseline and Day 84
Population: Intent-to-Treat (ITT) Population: all randomized participants who received at least 1 dose of randomized study drug in the Treatment Period. Participants analyzed were those with data available at the presented time point; but, all participants without missing covariate information and with >= post BL measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 mcg | FSC 250/50 mcg
Number analyzed (Participants) | 349 | 348
Liters | 0.213 (0.0137) | 0.112 (0.0139)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg vs FSC 250/50 mcg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.063 to 0.139] — Least squares mean difference=UMEC/VI 62.5/25 mcg minus FSC 250/50 mcg

2. Secondary Outcome: Change From Baseline(BL) in Trough Forced Expiratory Volume in One Second (FEV1) at Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Baseline is defined as the mean of the assessments made 30 and 5 minutes (min) pre-dose on treatment Day 1. Trough FEV1 on Day 85 is defined as the mean of the FEV1 values obtained 23 and 24 hours after morning dosing on Day 84. Analysis was performed using a repeated measures model with covariates of treatment, Baseline (mean of the 2 assessments made 30 min and 5 min pre-dose on Day 1), smoking status, day, day by baseline and day by treatment interactions. The model used all available trough FEV1 values recorded on Days 28, 56, 84, and 85. Missing data were not directly imputed in this analysis; however, all non-missing data for a participant were used within the analysis to estimate the treatment effect for trough FEV1 at Day 85. Change from baseline was calculated as the value at Day 84 minus the value at Baseline.
Time Frame: Baseline and Day 85
Population: ITT Population. Participants analyzed were those with data available at the presented time point; but, all participants without missing covariate information were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 mcg | FSC 250/50 mcg
Number analyzed (Participants) | 349 | 348
Liters | 0.185 (0.0138) | 0.087 (0.0140)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) collected from the start of study treatment up to the Follow-up Visit or premature withdrawal (up to Day 94)
Description: SAEs and non-serious AEs are reported for members of the ITT Population,comprised of all randomized participants who received at least 1 dose of randomized study drug in the treatment period
Arm/Group | UMEC/VI 62.5/25 mcg | FSC 250/50 mcg
Serious Adverse Events (participants affected / at risk) | 11/349 | 13/348
Other Adverse Events (participants affected / at risk) | 36/349 | 28/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 mcg (N=349) | FSC 250/50 mcg (N=348)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4
Appendicitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 mcg (N=349) | FSC 250/50 mcg (N=348)
Headache (Nervous system disorders) | 24 | 23
Nasopharyngitis (Infections and infestations) | 14 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.